CLINICAL TRIAL: NCT00965523
Title: Phase II Extension Study of E7389 for Locally Advanced or Metastatic Breast Cancer
Brief Title: Study of E7389 for Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-J081-224; E7389-J081-221; NCT00633100 (obsolete NCT alias)
Record Dates: First submitted 2009-08-20; First posted 2009-08-25 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2013-08-15 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Cancer; breast cancer; neoplasm; E7389; Eribulin
MeSH Terms: conditions — Breast Neoplasms; Neoplasms | interventions — eribulin

ARMS (1):
- Eribulin Mesylate (Experimental)
  Interventions: Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Eribulin Mesylate — Eribulin mesylate 1.4 mg/m^2 intravenous infusion (IV) given over 2 to 5 minutes on Day 1 and 8 every 21 days.

SUMMARY:
The purpose of this study (E7389-J081-224; hereafter referred to as Study 224) is to evaluate the safety of patients who continue to receive E7389 after completing the Phase II clinical study (E7389-J081-221; hereafter referred to as Study 221) of E7389 for advanced or relapsed breast cancer by intravenously administering E7389.

DETAILED DESCRIPTION:
Study 224 (Extension Period) was designed to evaluate the safety and efficacy of E7389 by collecting data from subjects who continued receiving E7389 after being transferred from Study 221 (Core Period). Thus, efficacy analyses performed in Study 221 were updated and reported with the additional data collected in Study 224. Objective response rate (ORR) and the number of subjects with adverse events are reported as outcome measures because these were the outcome measures of Study 221 which is a main study in the combined data. Also, safety analyses performed in Study 221 were updated and reported with the additional data collected in Study 224.

ELIGIBILITY:
Inclusion criteria:

1. Female patients with histologically or cytologically confirmed breast cancer.
2. Patients who have received prior chemotherapy including anthracycline and taxane.
3. Patients aged 20 - 74 years when giving informed consent and who have given written voluntary consent for participating in this study before the completion of Study 221.
4. Patients with an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 to 2.
5. Patients with a measurable lesion.
6. Patients with an expected survival of ≥ 3 months from the start of study drug therapy.
7. Female patients in whom continued administration of E7389 following Study 221 will be useful.
8. Patients who have met the criteria for starting the next cycle in Study 221.

Namely, patients who meet all of the following criteria:

1. Neutrophil count >= 1,500 /µL
2. Platelet count >= 100,000 /µL
3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 times the upper limit of normal (ULN) in the facility or <= 5 times ULN in patients with hepatic metastasis)
4. Total bilirubin <= 1.5 times ULN
5. Serum creatinine <= 1.5 times ULN
6. Non-hematological toxicity <= Grade 2 (excluding disease-associated events and laboratory abnormalities without clinical symptoms)

Exclusion criteria:

1. Patients with systemic infection with a fever (≥38.0°C).
2. Patients with pleural effusion, ascites or pericardial fluid requiring drainage.
3. Patients with brain metastasis presenting clinical symptoms.
4. Pregnant women, nursing mothers, or premenopausal women of childbearing potential. Premenopausal women of childbearing potential are defined as women who are <12 months after the latest menstruation and are positive in pregnancy test performed for enrollment or who have not taken the test and do not consent to take an appropriate contraceptive measure. Post-menopausal women must be amenorrheic for at least 12 months to make sure that they have no potential for becoming pregnant.
5. Patients with serious complications:

   1. Patients with uncontrollable cardiac disease such as ischemic heart disease and arrhythmia at a level of severity that needs to be treated (excluding left ventricular hypertrophy, mild left ventricular volume overload and mild right leg block that accompany hypertension)
   2. Patients with myocardial infarction within 6 months prior to study entry
   3. Patients with a complication of hepatic cirrhosis
   4. Patients with interstitial pneumonia and pulmonary fibrosis
   5. Patients with a bleeding tendency
6. Patients with an active double cancer.
7. Pregnant women or nursing mothers.
8. Patients who have received extensive radiotherapy (≥30% of bone marrow).
9. Patients who refuse to receive the supportive therapy of blood transfusion for myelosuppression.
10. Patients who are participating in other clinical studies.
11. Patients who are judged by the principal investigator or the other investigators to be inappropriate as patients in this clinical study.

Ages: 20 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-01; Primary Completion 2010-12 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tatsuo Watanabe, Study Director — Oncology Clinical Development Section. JAC PCU., Eisai, Co., Ltd
Locations (5):
- Japan (5):
  - Nagoya, Aichi-ken
  - Fukuoka, Fukuoka
  - Kure, Hiroshima
  - Kagoshima, Kagoshima-ken
  - Chūō, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study 221 was conducted at 22 centers in Japan during the period of Jan 2008 to Sept 2009, and Study 224 was conducted at 5 centers in Japan from Aug 2009 to Jan 2011.
Pre-assignment Details: Study 224 was designed to evaluate the safety and efficacy of E7389 by collecting data from subjects who continued receiving E7389 after being transferred from Study 221. Thus, combined data of Study 221 and Study 224 are reported.
Groups:
- Eribulin Mesylate: Eribulin mesylate 1.4 mg/m^2 intravenous infusion given over 2 to 5 minutes on Day 1 and 8 every 21 days.
Period: Study 221
Arm/Group | Eribulin Mesylate
Started | 81 (Study 221 (Safety Analysis Set).)
Completed | 74
Not Completed | 7
Not completed — Progressive Disease | 4
Not completed — Physician Decision | 3
Period: Study 224
Arm/Group | Eribulin Mesylate
Started | 6 (Six subjects continued into Study 224 from Study 221.)
Completed | 0
Not Completed | 6
Not completed — Progressive Disease | 5
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Demographic data were reported for 80 subjects, the Full Analysis Set, which is the primary efficacy analysis set in this study.
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 80
Age Continuous [Mean (Standard Deviation); unit: years] | 53.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80
  Male | 0
Region of Enrollment [Number; unit: participants] — Full Analysis Set
  participants
    Japan | 80

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Events.
Time Frame: Every week during treatment and up to 30 days after last dose of study treatment
Population: Safety Analysis Set
Measure: Number; unit: Participants
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 81
Participants | 81

2. Secondary Outcome: Objective Response Rate (ORR) as Measured by Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Objective response measured by Response Evaluation Criteria In Solid Tumors (RECIST) criteria and is Complete Response (disappearance of all target lesions) plus Partial Response (at least 30% decrease in sum of longest diameter [LD] of target lesions compared baseline sum of LD). Tumor assessments every 6 weeks.
Time Frame: Every 6 weeks
Population: Full Analysis Set
Measure: Number; unit: percentage of subjects
Arm/Group | Eribulin Mesylate
Number analyzed (Participants) | 80
percentage of subjects
  Objective Response Rate | 21.3 [29 to 431]
  Partial Response | 21.3
  Stable Disease | 37.5
  Progressive Disease | 40.0
  Not Evaluable | 1.3

ADVERSE EVENTS:
Arm/Group | Eribulin Mesylate
Serious Adverse Events (participants affected / at risk) | 14/81
Other Adverse Events (participants affected / at risk) | 81/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=81)
Neutropenia (Blood and lymphatic system disorders) | 1
Cataract (Eye disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Gastritis Hemorrhagic (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stomatitis (Gastrointestinal disorders) | 2
Malaise (General disorders) | 1
Oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Infection (Infections and infestations) | 2
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcemia (Metabolism and nutrition disorders) | 1
Decreased Appetite (Metabolism and nutrition disorders) | 2
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 1
Hemorrhage (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eribulin Mesylate (N=81)
Febrile Neutropenia (Blood and lymphatic system disorders) | 12
Leukopenia (Blood and lymphatic system disorders) | 80
Lymphopenia (Blood and lymphatic system disorders) | 44
Neutropenia (Blood and lymphatic system disorders) | 80
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Constipation (Gastrointestinal disorders) | 14
Diarrhea (Gastrointestinal disorders) | 15
Nausea (Gastrointestinal disorders) | 36
Stomatitis (Gastrointestinal disorders) | 33
Vomiting (Gastrointestinal disorders) | 16
Abdominal Pain Upper (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 37
Malaise (General disorders) | 11
Pain (General disorders) | 9
Pyrexia (General disorders) | 25
Chest Pain (General disorders) | 5
Oedema (General disorders) | 7
Nasopharyngitis (Infections and infestations) | 22
Infection (Infections and infestations) | 6
Alanine Aminotransferase Increased (Investigations) | 27
Aspartate Aminotransferase Increased (Investigations) | 30
Blood Albumin Decreased (Investigations) | 10
Blood Creatine Phophokinase Increased (Investigations) | 23
Blood Glucose Increased (Investigations) | 12
Blood Lactate Dehydrogenase Increased (Investigations) | 16
C-Reactive Protein Increased (Investigations) | 14
Gamma Glutamyltransferase Increased (Investigations) | 22
Blood Urine Present (Investigations) | 8
Hemoglobin Decreased (Investigations) | 28
Weight Decreased (Investigations) | 9
Blood Alkaline Phosphatase Increased (Investigations) | 18
Red Blood Cell Count Decreased (Investigations) | 5
Decreased Appetite (Metabolism and nutrition disorders) | 38
Hyperglycemia (Metabolism and nutrition disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 14
Back Pain (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 8
Dizziness (Nervous system disorders) | 9
Dysgeusia (Nervous system disorders) | 27
Headache (Nervous system disorders) | 13
Peripheral Sensory Neuropathy (Nervous system disorders) | 19
Hypoaesthesia (Nervous system disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 8
Alopecia (Skin and subcutaneous tissue disorders) | 47
Rash (Skin and subcutaneous tissue disorders) | 11
Anemia (Blood and lymphatic system disorders) | 7
Oedema Peripheral (General disorders) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No